CLINICAL TRIAL: NCT07211555
Title: The LARC Robot Simplifies Renal Access In Percutaneous Nephrolithotomy (PCNL)
Brief Title: The LARC Robot Simplifies Renal Access In Percutaneous Nephrolithotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2196760
Record Dates: First submitted 2025-07-16; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-07

CONDITIONS: Renal Stone Disease; Kidney Calculi; Refractory Kidney Stones; Kidney Stones
Keywords: Robotic Surgery; Minimally Invasive Surgery
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Assisted PCNL Using LARC System (Experimental): This arm includes participants who will undergo percutaneous nephrolithotomy (PCNL) with renal access guided by the investigational LARC robotic system (Version 3.0). The procedure uses fluoroscopy-based navigation to assist the urologist in targeting the renal collecting system.
  Interventions: Device: LARC Robotic System (Micromate™ Version 3.0)

INTERVENTIONS:
Device: LARC Robotic System (Micromate™ Version 3.0) — The LARC Robotic System (Version 3.0) is an investigational configuration of the Micromate™ robotic platform by iSYS Medizintechnik GmbH (Austria). It uses fluoroscopy-based surgical navigation to assist urologists in obtaining precise renal access during percutaneous nephrolithotomy (PCNL). This version is not FDA-cleared and is being evaluated for feasibility, safety, and potential clinical benefit.

SUMMARY:
This study is being done to evaluate a new robotic system that helps urologists more precisely reach the kidney during surgery to remove large kidney stones. The procedure, called percutaneous nephrolithotomy (PCNL), is typically used for people who have large or difficult-to-remove kidney stones.

Traditionally, many urologists rely on radiologists to place a tube into the kidney before surgery. This can cause delays, require multiple procedures, and increase costs. The robotic system being studied - called LARC - is designed to help the urologist safely and accurately guide a needle directly into the kidney during the surgery, without needing a separate procedure beforehand.

The robot uses live X-ray images to help align the instruments. Although parts of the robot have been approved by the U.S. FDA, the version used in this study is still investigational and not yet approved for this specific purpose.

The study will take place at AdventHealth Celebration and include up to 45 adult patients who are scheduled for PCNL surgery. Participants will be followed for up to 1 month after surgery, and doctors will look at outcomes such as the success of the procedure, the number of kidney stones removed, complications, time in surgery, and radiation exposure.

This research may help make kidney stone surgery safer, faster, and more effective in the future.

ELIGIBILITY:
Inclusion Criteria:

* Kidney stones larger than 2 cm
* Staghorn renal calculi
* Lower pole stones less than 2 cm
* Anatomical abnormalities that reduce the likelihood of spontaneous stone fragment passage, such as:
* Horseshoe kidney
* Calyceal diverticulum
* Ectopic or dystopic kidney
* Stones that are refractory to prior treatment (e.g., ESWL or ureteroscopy)
* Suspected malignant tumors or masses located in the planned renal access tract

Exclusion Criteria:

* Pregnancy
* Active urinary tract infection (UTI) or untreated sepsis
* Known bleeding disorders or uncorrectable coagulopathy despite medical management
* Use of anticoagulant medications (e.g., warfarin, heparin, or DOACs) that cannot be safely discontinued
* Allergy to contrast media that cannot be pre-medicated or managed
* Severe cardiopulmonary comorbidities that contraindicate anesthesia or PCNL
* Inability to provide informed consent
* Participation in another investigational study that may interfere with study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Stone-Free Rate (SFR) | Within 30 days post-procedure
  Proportion of participants with no residual kidney stones larger than 4 mm, as determined by imaging (non-contrast CT, KUB X-ray, or renal ultrasound).
Procedure Success Rate | During procedure (Day 0)
  Proportion of procedures in which the urologist was able to successfully obtain renal access and complete the PCNL using the LARC robotic system, without converting to manual or radiologist-assisted access.

SECONDARY OUTCOMES:
Estimated Blood Loss (EBL) | During procedure (Day 0)
  Volume of blood loss (in mL) recorded during PCNL using the LARC system, measured via standard intraoperative methods.
Operative Time | During procedure (Day 0)
  Total time (in minutes) from skin incision to procedure completion. Sub-analysis includes time from renal access start to access success.
Radiation Exposure | During procedure (Day 0)
  Total fluoroscopy time and radiation dose (in mGy and seconds) recorded during robotic-assisted access using the LARC system.
Postoperative Complications | Up to 30 days post-procedure
  All adverse events will be recorded and graded using the Clavien-Dindo classification system. Includes infection, transfusion, organ injury, and reintervention.
Number of Access Attempts | During procedure (Day 0)
  Number of needle punctures required to achieve access to the renal collecting system.

CONTACTS AND LOCATIONS:
Locations (1):
- Advent Health Medical Group Urology at Celebration, Celebration, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing information from this study.

REFERENCES:
- [Background] Escobar Monroy R, Proietti S, De Leonardis F, Gisone S, Scalia R, Mongelli L, Gaboardi F, Giusti G. Complications in Percutaneous Nephrolithotomy. Complications. 2025; 2(1):5. https://doi.org/10.3390/complications2010005
- [Background] Nguyen MV, Berger JH, Flores AR, Chen TT, Yared J, Pais V, Chew B, Humphreys MR, Stern KL, Sur RL. Case series - Liver injury during percutaneous nephrolithotomy. Can Urol Assoc J. 2023 Sep;17(9):E297-E301. doi: 10.5489/cuaj.8291. No abstract available. PMID 37458736
- [Background] Saluk J, Ebel J, Rose J, Posid T, Sourial M, Knudsen B. Fellowship training in endourology: Impact on percutaneous nephrolithotomy access patterns. Can Urol Assoc J. 2022 Feb;16(2):E76-E81. doi: 10.5489/cuaj.7339. PMID 34582338
- [Background] Taylor E, Miller J, Chi T, Stoller ML. Complications associated with percutaneous nephrolithotomy. Transl Androl Urol. 2012 Dec;1(4):223-8. doi: 10.3978/j.issn.2223-4683.2012.12.01. No abstract available. PMID 26816715
- [Background] de la Rosette J, Assimos D, Desai M, Gutierrez J, Lingeman J, Scarpa R, Tefekli A; CROES PCNL Study Group. The Clinical Research Office of the Endourological Society Percutaneous Nephrolithotomy Global Study: indications, complications, and outcomes in 5803 patients. J Endourol. 2011 Jan;25(1):11-7. doi: 10.1089/end.2010.0424. PMID 21247286
- [Background] Korets R, Speed JM, Wang Y, Chang SL. PD21-03 Percutaneous Access Obtained By Urologist Is Associated With Decreased Complications, Shorter Length Of Stay, And Lower Hospital Costs In PCNL. J Urol. 2017;197(4S):e436-e437. doi:10.1016/j.juro.2017.02.1041
- [Background] Ghoulian J, Nourian A, Dalimov Z, Ghiraldi EM, Friedlander JI. Percutaneous Nephrolithotomy Access: A Meta-Analysis Comparing Access by Urologist vs Radiologist. J Endourol. 2023 Jan;37(1):8-14. doi: 10.1089/end.2022.0308. Epub 2022 Nov 14. PMID 36136905
- [Background] Armitage JN, Withington J, Fowler S, Finch WJG, Burgess NA, Irving SO, Glass J, Wiseman OJ; BAUS section of Endourology. Percutaneous nephrolithotomy access by urologist or interventional radiologist: practice and outcomes in the UK. BJU Int. 2017 Jun;119(6):913-918. doi: 10.1111/bju.13817. Epub 2017 Mar 21. PMID 28220589
- [Background] Speed JM, Wang Y, Leow JJ, Bhojani N, Trinh QD, Chang SL, Korets R. The Effect of Physician Specialty Obtaining Access for Percutaneous Nephrolithotomy on Perioperative Costs and Outcomes. J Endourol. 2017 Nov;31(11):1152-1156. doi: 10.1089/end.2017.0441. Epub 2017 Oct 4. PMID 28859496
- [Background] Quirke K, Aydin A, Brunckhorst O, Bultitude M, Khan MS, Dasgupta P, Sarica K, Ahmed K. Learning Curves in Urolithiasis Surgery: A Systematic Review. J Endourol. 2018 Nov;32(11):1008-1020. doi: 10.1089/end.2018.0425. PMID 30039711
- [Background] Metzler IS, Holt S, Harper JD. Surgical Trends in Nephrolithiasis: Increasing De Novo Renal Access by Urologists for Percutaneous Nephrolithotomy. J Endourol. 2021 Jun;35(6):769-774. doi: 10.1089/end.2020.0888. Epub 2021 Apr 5. PMID 33430693